CLINICAL TRIAL: NCT04366232
Title: Interleukin-1 (IL-1) and Interferon Gamma (IFNg) Inhibition During COVID 19 Inflammation: Randomized, Controlled Study Assessing Efficacy and Safety of Anakinra and Ruxolitinib
Brief Title: Efficacy of Intravenous Anakinra and Ruxolitinib During COVID-19 Inflammation
Acronym: JAKINCOV
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: investigator decision
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Hôpital d'instruction des armées Sainte-Anne (Unknown); Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-CHITS-003; 2020-001963-10 (EudraCT Number)
Record Dates: First submitted 2020-04-27; First posted 2020-04-28 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Covid-19
Keywords: COVID; SARS-CoV-2; Anakinra; Ruxolitinib; IL-1 inhibitors; JAK inhibitors
MeSH Terms: conditions — COVID-19 | interventions — Interleukin 1 Receptor Antagonist Protein; ruxolitinib; Standard of Care

STUDY DESIGN:
Intervention Model Description: Assignment to one of two or more groups in parallel during the study No crossover
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anakinra +/- Ruxolitinib (Experimental): According to clinical stage (gradual strategy):
  * Stage 2b or 3 : Anakinra 300 mg IV
  * Overcome stage 3 : Anakinra 300 mg IV and Ruxolitinib 5 mg x 2
  Interventions: Drug: Anakinra alone (stages 2b/3); Drug: Anakinra and Ruxolitinib (overcome stage 3)
- Standard of care (Active Comparator): Treatment with drugs or procedures in routine clinical practice
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Anakinra alone (stages 2b/3) — Anakinra 300 mg 1/d Intravenous 5 days then dose tapering
  Other Names: KINERET
  Arms: Anakinra +/- Ruxolitinib
Drug: Anakinra and Ruxolitinib (overcome stage 3) — Anakinra 300 mg od Intravenous (maximum14 days) Ruxolitinib 5 mg bid per os (maximum 28 days)
  Other Names: KINERET and JAKAVI
  Arms: Anakinra +/- Ruxolitinib
Other: Standard of care — Routine clinical care for Covid-19
  Arms: Standard of care

SUMMARY:
During SARS-Cov2 infection with serious respiratory implication and high systemic inflammation level, intravenous ANAKINRA alone or associated with RUXOLITINIB for severe cases might reduce inappropriate systemic inflammatory response, improve breathing and decrease occurrence or duration of ARDS and associated mortality.

DETAILED DESCRIPTION:
Two physiopathological phases exist during COVID-19 disease: The early phase is mainly induced by the virus itself. It is imperative not to decrease the immune host response during this phase by prohibiting the use of non steroidal anti-inflammatory drugs or corticosteroids at this stage and developing an anti-viral strategy. The late phase, around Day 7-9, depends only upon host response and is linked to an excessive inflammatory response with a major increase of inflammatory cytokines such as IL-6, MCP-1, GCSF indicative of IL-1b excess, as well as IP-10, MIP-1, indicative of IFNg signature, corresponding to a "cytokine storm". Clinical and biological features during Still's disease (complicated in 10% of cases with hemophagocytosic lymphohistiocytosis inducing cytopenia, hepatic insufficiency, major hyperferritinemia and multi-organ failure) are close to those reported during COVID-19 and underline physiopathological similarities.

Anakinra (KINERET) is an IL-1 pathway (IL-1ra) specific inhibitor that has been used for 15 years, also largely blocking IL-18 production. Adult Still's disease is very effectively treated with anakinra. During sepsis with hyperferritinemia, IL-1ra demonstrated patient survival improvement. Ruxolitinib (JAKAVI) inhibits the downstream IFNg pathway targeting JAK kinase receptor. It has recently proved its efficiency in hemophagocytosic lymphohistiocytosis refractory forms associated with a multi-organ failure.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed respiratory tract SARS-coV-2 infection by at least one PCR on nasopharygeal sample or a bronchoalveolar lavage
* Patient hospitalized with clinical, biological and radiological features corresponding to the following stages :

  * Stage 2b: hypoxic pneumonia (respiratory frequency > 30/mn, Sa02 < 90 mmHg on room air) associated with a clear biological inflammatory syndrome (CRP > 150 mg/l)
  * Stage 3: ARDS defined by a patient under mechanical ventilation with a ratio PaO2/FiO2 < 300 for more than 24h
  * Evolved stage 3: ARDS according to previous definition associated with another organ failure or syndrome among:
* A state of shock with noradrenaline dosing > 3mg/h
* Acute kidney failure oligo-anuric or justifying extra-renal purification
* Hepatocellular insufficiency or coagulopathy with a V factor < 50%
* Myocarditis responsible for acute heart failure and or cardiogenic shock
* Hemophagocytic syndrome
* Hyperferritinemia > 5000 ng/mL
* Subject or legal representative having expressed written consent after information
* Subject affiliated to or entitled to a social security regimen
* Patient presenting in a life-threatening emergency situation that does not allow consent to be obtained

Exclusion Criteria:

* Pregnancy or lactation
* Absolute neutrophil count less than 1.5 x 109/L
* Hepatic transaminases AST or ALT greater than 5 times normal values
* Platelet count less than 50,000 per mm3
* Solid organ or hematopoietic stem cell transplant patients
* Patients treated with immunosuppressants or immunomodulators
* Use of oral corticosteroids chronically at doses greater than 10 mg prednisone equivalent per day for a non-COVID-19 related condition.
* Uncontrolled autoimmune disease
* Patients with active, suspected or known, uncontrolled systemic bacterial, viral (excluding COVID-19) or fungal infections
* Hypersensitivity to anakinra and/or ruxolitinib and their excipients
* Vaccinations with live attenuated vaccines in the month prior to inclusion
* Patients with severe pre-existing uncontrolled organ dysfunction (heart, liver or kidney failure)
* Persons deprived of liberty by judicial or administrative decision or major persons under a legal protection measure.
* Person in exclusion period of another research protocol for SARS-CoV-2 infection.
* Person not mastering enough French understanding and reading to be able to consent to participate in the study.
* Persons under psychiatric care pursuant to Articles A3112-1 and L3113-1 who are not covered by the provisions of Article L1121-8
* Every condition which, according to investigator, might increase and compromise the person security in case of study participation or might interfere with research results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Biological criteria | 7 days from enrolment
  At least 3 parameters are met including CRP and/or Ferritin among:
  1. CRP: decrease > 50%
  2. Ferritinemia: decrease > 1/3
  3. Serum creatinine: decrease > 1/3
  4. AST/ALT: decrease > 50%
  5. Eosinophils > 50 /mm3
  6. Lymphocytes > 1000 /mm3

SECONDARY OUTCOMES:
Duration of oxygen therapy (days) | 28 days from enrolment
  Number of days without mechanical ventilation
Number of intensive care units admissions | 28 days from enrolment
  Number of patients included in stage 2b
Number of days in intensive care units | 28 days from enrolment
  Number of days in intensive care units for patients managed in intensive care units
Mortality rate | 28 days from enrolment
  Mortality rate
Total number of days in hospital | 28 days from enrolment
  Total number of days in hospital
Organ failure score modification (Sepsis-related Organ Failure Assessment (SOFA) score) | 28 days from enrolment
  Organ failure score modification (Sepsis-related Organ Failure Assessment (SOFA) score); Sofa score's minimum and maximum values are 0 and 24, the lowest score corresponds to a better outcome.
Number of bacterial and/or fungal sepsis | 28 days from enrolment
  Number of bacterial and/or fungal sepsis

CONTACTS AND LOCATIONS:
Overall Officials: David DELARBRE, MD, Principal Investigator — French Army Health Service
Locations (3):
- France (3):
  - AP-HM, Hôpital de la Conception, Marseille, Bouches-du-Rhône
  - Hôpital Sainte-Musse, Toulon, VAR
  - Sainte Anne Teaching Military Hospital, Toulon, Var

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Zalinger ZB, Elliott R, Weiss SR. Role of the inflammasome-related cytokines Il-1 and Il-18 during infection with murine coronavirus. J Neurovirol. 2017 Dec;23(6):845-854. doi: 10.1007/s13365-017-0574-4. Epub 2017 Sep 11. PMID 28895072